CLINICAL TRIAL: NCT00001176
Title: The Function of Dopaminergic and Noradrenergic Systems in Salt-Sensitive Hypertension: The Effects of Changes in Sodium Intake
Brief Title: Effects of Salt Intake on the Nervous Systems of Patients With Salt-Sensitive High Blood Pressure
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 810081; 81-H-0081
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-12

CONDITIONS: Hyperaldosteronism; Hypertension
Keywords: Adrenergic Nervous System; Dopaminergic Nervous System; Salt-Sensitive Hypertension; Hypertension; Primary Aldosteronism
MeSH Terms: conditions — Hyperaldosteronism; Hypertension

SUMMARY:
Some patients with high blood pressure can experience an increase of blood pressure by 10 percent or more by taking in salt. These patients are referred to as having "salt-sensitive" (SS) hypertension.

Previous studies conducted on patients with salt sensitive hypertension suggest that their portion of the nervous system responsible for maintaining normal blood pressure (autonomic nervous system) may respond differently to salt than patients with non-salt sensitive (NSS) hypertension.

This study is designed to examine the response of the nervous system to high doses of salt in patients with salt-sensitive hypertension and patients with non-salt sensitive hypertension.

DETAILED DESCRIPTION:
A subset of patients with idiopathic hypertension shows an increase in blood pressure of 10 percent or more in response to salt-loading and have been termed "salt-sensitive" (SS). Limited studies of adrenergic function in response to salt-loading suggest that the response of SS patients may differ from that of non-salt sensitive (NSS) patients. The present studies were designed to examine the response of the adrenergic and dopaminergic systems to salt-loading in SS and NSS patients with idiopathic hypertension.

ELIGIBILITY:
Eligibility criteria not identified in protocol.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110
Dates: Start 1981-05; Study Completion 2001-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kawasaki T, Delea CS, Bartter FC, Smith H. The effect of high-sodium and low-sodium intakes on blood pressure and other related variables in human subjects with idiopathic hypertension. Am J Med. 1978 Feb;64(2):193-8. doi: 10.1016/0002-9343(78)90045-1. PMID 629267
- [Background] Fujita T, Henry WL, Bartter FC, Lake CR, Delea CS. Factors influencing blood pressure in salt-sensitive patients with hypertension. Am J Med. 1980 Sep;69(3):334-44. doi: 10.1016/0002-9343(80)90002-9. No abstract available. PMID 6998291
- [Background] Alexander RW, Gill JR Jr, Yamabe H, Lovenberg W, Keiser HR. Effects of dietary sodium and of acute saline infusion on the interrelationship between dopamine excretion and adrenergic activity in man. J Clin Invest. 1974 Jul;54(1):194-200. doi: 10.1172/JCI107743. PMID 4600048